CLINICAL TRIAL: NCT03771209
Title: The "ABCDE" Score as a Five-step Vascular Ultrasound Examination in Heart Failure:a Multi-center Study
Brief Title: The "ABCDE" Score as a Five-step Vascular Ultrasound Examination in Heart Failure
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Azienda Ospedaliera Universitaria Integrata Verona (Other)
Collaborators: University of Palermo (Other); University Of Perugia (Other); IRCCS Sacro Cuore Don Calabria di Negrar (Other)
Responsible Party: Principal Investigator, Chiara Mozzini, Principal Investigator, Azienda Ospedaliera Universitaria Integrata Verona
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: ABCDE
Record Dates: First submitted 2018-12-05; First posted 2018-12-11 (Actual); Last update posted 2018-12-11 (Actual); Status verified 2018-12

CONDITIONS: Heart Failure; Atherosclerosis
Keywords: ultrasound assessment; ankle brachial index; lung ultrasound; carotid intima media thickness; vascular ultrasound (abdominal aorta and cave vein); echocardiographic ejection fraction
MeSH Terms: conditions — Heart Failure; Atherosclerosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- ultrasound assessment (Experimental): The aim of this study is the creation of a five-step ultrasound examination to evaluate and monitor HF patients during hospitalization and short follow-up.
  Interventions: Diagnostic Test: ultrasound examination

INTERVENTIONS:
Diagnostic Test: ultrasound examination — ultrasound assessment

SUMMARY:
Heart failure (HF) is a clinical syndrome caused by structural and/or functional cardiac abnormalities, resulting in a reduced cardiac output and/or elevated intra-cardiac pressures at rest or during stress. It is the leading cause of hospitalization in Internal Medicine departments.

This study aims at exploring evidence of the importance of ultrasound in HF both for hospitalized patients and in the follow up. Ultrasound may be used as a recovery monitoring instrument at the bedside and also as a global cardiovascular assessment tool for these patients.

HF represents an exciting opportunity to create an integrative ultrasound approach in Internal Medicine/Geriatric departments.The Authors plan a five-step ultrasound examination to evaluate and monitor HF patients during hospitalization and follow-up. They call this examination: the "ABCDE" score. It includes the evaluations of A, the Ankle-brachial index (ABI), B, the B-lines, C, the Carotid intima media thickness (CIMT), D, the Diameter of the abdominal aorta and of the inferior cave vein and E, the echocardiographic assessment of the ejection fraction.This score represent an integrative ultrasound approach in Internal Medicine/Geriatric departments.

DETAILED DESCRIPTION:
Background: Heart failure (HF) is a clinical syndrome characterized by typical symptoms and signs caused by structural and/or functional cardiac abnormalities, resulting in a reduced cardiac output and/or elevated intra-cardiac pressures at rest or during stress. The prevalence of HF is approximately 1-2% of the adult population in developed countries, rising to ≥10% among people >70 years of age and it is the leading cause of hospitalization.

The aim of this study is the creation of a five-step ultrasound examination to evaluate and monitor HF patients during hospitalization and short follow-up.

The "ABCDE" score includes the evaluations of A, the Ankle-brachial index, ABI, B, the B-lines, C, the Carotid intima media thickness, CIMT, D, the Diameter of the abdominal aorta and of the inferior cave vein and E, the echocardiographic assessment of the ejection fraction.

This score represents an integrative ultrasound approach in the Internal Medicine/Geriatric departments:

A (ANKLE-BRACHIAL INDEX) Normal (<90): points 0 Mild obstruction (0.71-0.90): points 1 Moderate obstruction (0.41-0.70): points 2 Severe obstruction 0-0.40): points 3 B (B-LINES) Number of B-lines for each space ≤5: points 0 Number of B-lines for each space ≥ 6 to ≤ 9: points 1 Number of B-lines for each space ≥ 10 ("Full white screen"): points 3 C (IMT OR CAROTID PLAQUE) Normal: points 0 Altered IMT (>0.9 mm): points 1 Plaque presence (no significant stenosis, <70% following NASCET classification): points 2 Plaque presence (significant stenosis, >70% following NASCET classification): points 3 D (DIAMETER OF AORTA AND VCI COLLAPSIBILITY INDEX) Aorta Normal (<25 mm): points 0 Normal diameter but with calcifications: points 1 Ectasia (25-30 mm): points 2 Aneurysm (>30mm): points 3 Cave Vein Normal collapsibility index (40-75%): points 0 Altered collapsibility index (if <40% or >75%): points 1 E (EF ACCORDING TO ESC GUIDELINES 2016) HFpEF (LVEF ≥50%): points 0 HFmrEF (LVEF in the range of 40-49%):points 1 HFrEF (LVEF<40%): points 2

Methods: The study population is composed of a consecutive sample of n' HF patients admitted from the Emergency to the Internal Medicine (IM)/Geriatric Departments of n' University Hospitals from Italy or other foreign countries.

HF criteria will be established according to the recent ESC 2016 guidelines. In particular, patients will be classified in three different classes: with normal left ventricular ejection fraction (LVEF) ( ≥50%, HF with preserved EF, HFpEF), with reduced LVEF ( <40%, HF with reduced EF, HfrEF) and with an LVEF in the range of 40-49% (HfmrEF).

Moreover, patients are classified according to New York Heart Association (NYHA) classes at admission, at discharge and during follow-up.

Exclusion criteria are: concomitant acute coronary syndrome, pneumonia, chronic obstructive pulmonary disease, lung cancer or metastases, lung fibrosis, previous pneumonectomy or lobectomy, breast prothesis, obesity, also in order to to avoid the detection of B-lines other than due to HF.

Patients undergo: A (calculated for each leg at admission), B-lines counting (calculated at admission, during hospital stay and at discharge with lung ultrasound, approach 72 spaces), C (at admission), D (at admission for the aorta and at admission, during hospital stay and at discharge for the inferior cave vein) and E (at admission and discharge).

Venous blood samples are collected from each subject for routine examination on admission: hemoglobin and white blood cells count, serum creatinine, sodium, potassium, urea, total cholesterol, high density lipoprotein (HDL) cholesterol, low density lipoprotein (LDL) cholesterol, triglycerides, glucose, C-reactive protein (CRP) (measured with standard methods).

Moreover, NT-proBNP dosage is obtained on admission and on discharge. Urine output and diuretic dosage will be carefully reported daily. Arterial blood samples is collected on admission and on discharge to test the partial pressure of oxygen (PaO2) as indicator of HF severity (on admission) and recovery (on discharge).

An electrocardiogram recording and X-chest ray examination are obtained on admission.

MEDICAL STAFF INVOLVED IN THE ULTRASOUND EXAMINATIONS A is performed by the IM/Geriatric specialists or certification board attending students.

B,C and D examinations are performed by Medical Doctors (Radiologists or IM/Geriatric specialists certified by the Società Italiana di Ultrasonologia in Medicina e Biologia (SIUMB).

Trans-thoracic echocardiography with estimation of E is performed by Cardiologists or IM specialists certified by the Società Italiana di Ecografia Cardiovascolare, SIEC.

* ENDPOINTS:

  1) RELATED TO THE BEDSIDE EVALUATION OF HF RECOVERY:
* test if B,D (for cave vein) and E assessment can precisely guide and tailoring the therapy (diuretics) during hospitalization and recovery from HF;
* test if B,D (for cave vein) and E assessment can speed up the discharge time (if compared to patients without ultrasound assessment);
* improve the use of bedside ultrasound in IM and Geriatric department. 2) RELATED TO THE GLOBAL CARDIOVASCULAR ASSESSMENT OF THE HF PATIENT:
* test if A, C and D (for aorta) assessment can better classify the global cardiovascular risk for the HF patient.

The severity of the score will be related with:

* number of hospitalization days
* number of "events" during follow up (for definition of "events", see follow up section).

FOLLOW-UP Follow-up is performed by contacting patients or their caregivers over the phone 30 and 90 days after the date of discharge. All the successive re-admissions for HF or deaths from any cause are considered as "events".

A potential correlation between the severity of each parameter considered in the "ABCDE" score with the "events" after discharge is tested.

ELIGIBILITY:
Inclusion Criteria:

* HF patients admitted from the Emergency to the Internal Medicine (IM)/Geriatric Departments

Exclusion Criteria:

* concomitant acute coronary syndrome
* pneumonia
* chronic obstructive pulmonary disease
* lung cancer or metastases
* lung fibrosis
* previous pneumonectomy or lobectomy
* breast prothesis
* obesity

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 480 (Estimated)
Dates: Start 2018-04-26 (Actual); Primary Completion 2022-04-26 (Estimated); Study Completion 2022-04-26 (Estimated)

PRIMARY OUTCOMES:
discharge time shortening | 1 month
  B-lines number in relation to the discharge time (number of days of hospitalization)
ABCDE and events | 3 months
  association between number of altered ultrasound parameters and number of "events" (death from any cause or re-admission for HF) in a follow up period (30 and 90 days from discharge)

SECONDARY OUTCOMES:
B lines and diuretics shifts | 1 month
  association between B lines number and the number of diuretics shifts during hospitalization and recovery from HF
B lines and PaO2 | 1 month
  association between B lines number and calculated ratio of arterial oxygen partial pressure to fractional inspired oxygen (PaO2/FiO2 ratio) at admission and discharge
B lines and natriuretic peptide | 1 month
  the association of B lines number and natriuretic peptide blood levels (ng/mL)

CONTACTS AND LOCATIONS:
Overall Officials: CHIARA MOZZINI, MD,PhD, Principal Investigator — Universita di Verona; DOMENICO GIRELLI, MD,PhD, Study Chair — Universita di Verona; MAURIZIO SORESI, MD,PhD, Study Chair — University of Palermo
Locations (1):
- University of Verona, Verona, Italy

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Mozzini C, Cominacini L, Casadei A, Schiavone C, Soresi M. Ultrasonography in Heart Failure: A Story that Matters. Curr Probl Cardiol. 2019 Apr;44(4):116-136. doi: 10.1016/j.cpcardiol.2018.05.003. Epub 2018 Jun 21. PMID 30172551